CLINICAL TRIAL: NCT00555529
Title: Systemic Endothelial Abnormalities in COPD Measured by Radial Artery Applanation Tonometry (RAAP)
Brief Title: Systemic Endothelial Abnormalities in COPD
Status: Withdrawn | Type: Observational
Why Stopped: Lead researcher left the Department
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 9022006
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exhaled breath condensate; applanation tonometry; induced sputum; smokers; healthy control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- 1
  Interventions: Procedure: radial artery applanation tonometry (RAAP)
- 2
  Interventions: Procedure: radial artery applanation tonometry (RAAP)

INTERVENTIONS:
Procedure: radial artery applanation tonometry (RAAP) — non-invasive tonometry

SUMMARY:
The purpose of this project is to validate the peripheral arterial pressure waveform measurements technique of RAAP (radial artery applanation tonometry), in patients with moderate and severe COPD (Chronic Obstructive Pulmonary Disease), and to assess the degree of systemic endothelial dysfunction in these patients compared to cigarette smokers with normal lung function and non-smokers with normal lung function.

DETAILED DESCRIPTION:
Patients with moderate and severe COPD (GOLD stage II and III) will be studied and their results will be compared with age-matched healthy non- smokers and smokers.

RAAP will be taken every 5 minutes for 15 minutes before salbutamol and every 5 minutes for another 15 minutes after salbutamol.

Several parameters of lipoprotein profiles, anti-oxidant plasma capacity, inflammatory cytokines, hormones, growth factors and vascular cell adhesion molecules will be studied in blood. In addition, several inflammatory and oxidative markers will be studied in exhaled breath condensate. Lung function and impulse oscillometry will be made to investigate airway resistance, and exhaled NO (nitric oxide) at different expiratory flows will be measured to assess alveolar and bronchial NO. Clinical assessment including dyspnoea and depression scores will also be made.

ELIGIBILITY:
Inclusion Criteria:

* • Male subjects with COPD with FEV1/FVC<70%; predicted defined as either stage moderate GOLD II (n=15) and severe GOLD III (n=7) diagnosis according to GOLD criteria (Global Strategy for the Diagnosis, Management, and Prevention of COPD) or Male subjects who are age-matched non-smokers (n=8) and male smokers (n=8) with normal lung function (FEV1>80%, FEV1/FVC>70%, n=8)

  * Smokers:

An active smoker with a pack history of >10 pack years [number of pack years = (number of cigarettes per day / 20) x number of years smoked]. Smokers need to report the time when last cigarette was smoked (no less than 6 hours before the study visit).

* Patients will be allowed to use their current anticholinergic bronchodilators and continue on the dose of inhaled corticosteroids they are currently using. However they should refrain from short and long-acting β2-agonists for 6 and 12 hours, respectively, before the study visit.
* Aged 40 80 years inclusive
* Body mass index within the range 19-32kg/m2 inclusive
* FEV1 <15% reversibility (not % predicted) and an increase of <200ml after inhaled β2-agonists (400μg salbutamol).
* Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject is available to complete the study.

Exclusion Criteria:

* • As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.

  * The subject has participated in a study with a new molecular entity during the previous 3 months or any other clinical trial during the previous 3 months. In case of a non invasive, clinical trial not involving new molecular entities a 2 week washout will be sufficient
  * The subject regularly, or on average, drinks more than 21 units of alcohol per week.
  * The subject has received oral steroids within 2 weeks prior to study entry.
  * The subject has history of an upper respiratory infection (including sinusitis) within 2 weeks prior to study entry
  * The subject has been hospitalised for a COPD exacerbation within 1 month of study entry.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers, COPD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01 (Estimated); Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London; Peter J Barnes, MD, Study Director — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial College London, London
  - National Heart and Lung Institute, London

REFERENCES:
- See also: Imperial College London — http://www3.imperial.ac.uk/